CLINICAL TRIAL: NCT02151123
Title: Metabiomics Colon Cancer Clinical Research Study
Status: Withdrawn | Type: Observational
Why Stopped: funding not secured
Sponsor: Metabiomics Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-02_CU
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2018-08

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; Colon Cancer; Microbiome
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gut microbiome samples from stool, rectal and colonic mucosa
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosed colon cancer patients: Patients undergoing colectomy for colonic adenocarcinoma.

SUMMARY:
The specific aim of the study is to determine the false negative rate of the Metabiomics Colon Polyp and Colorectal Cancer Assay for Cancer.

DETAILED DESCRIPTION:
The purpose of this study is to conduct clinical research to investigate the association of the gut microbiome with colonic neoplasia. In this case several types of gut microbiome samples will be collected from patients undergoing colectomy for colonic adenocarcinoma; those samples will be tested by Metabiomics Colon Polyp and Colorectal Cancer Assay and the percentage of false negative (test returns a negative for cancer) results determined.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with colorectal cancer (CRC) and scheduled for colectomy
* Male or female,
* Age: 18-95 years,
* Able to comprehend, sign, and date the written informed consent form (ICF),
* Able to give informed consent in English
* Women and minorities will be included.

Exclusion Criteria:

* History of Inflammatory Bowel Disease
* Antibiotics within 2 weeks of sample collection.
* Colonoscopy, colon prep or bowel contrast agent within 7 days prior to sample collection
* Any radiation therapy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colonic adenocarcinoma undergoing colectomy at University of Colorado
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
False negative rate of test for colon cancer | immediately post surgery
  The False Negative Rate is calculated as (100*False Negative) /(True Positive + False Negative).

CONTACTS AND LOCATIONS:
Overall Officials: Jon Vogel, MD, Principal Investigator — University of Colorado School of Medicine Anschutz Medical Campus; Christopher Lieu, MD, Principal Investigator — University of Colorado School of Medicine Anschutz Medical Campus; Patrick Gillevet, PhD, Principal Investigator — George Mason University
Locations (1):
- University of Colorado School of Medicine Anschutz Medical Campus, Aurora, Colorado, United States